CLINICAL TRIAL: NCT07133230
Title: Neurocognitive Correlates of the Influence of Number Word Syntax on Magnitude Processing
Acronym: NUMWORD
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D24-P010
Record Dates: First submitted 2025-06-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-05

CONDITIONS: Brain Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants recruited (phase 1): In each experimental phase (2 in total), 42 adult volunteers will be recruited (a total of 84 participants), selected based on the following criteria:
  * Aged 18-45
  * Female or male
  * Right-handed
  * Signed informed consent
  * Normal medical, neurological, and neuroradiological examinations
  * Affiliated with a social security system
  * For women of childbearing age: under effective contraception; a urine pregnancy test will be administered
  * MRI examination compatible Participants will be recruited in the Paris region.
- Participants recruited (phase 2): In each experimental phase (2 in total), 42 adult volunteers will be recruited (a total of 84 participants), selected based on the following criteria:
  * Aged 18-45
  * Female or male
  * Right-handed
  * Signed informed consent
  * Normal medical, neurological, and neuroradiological examinations
  * Affiliated with a social security system
  * For women of childbearing age: under effective contraception; a urine pregnancy test will be administered
  * MRI examination compatible Participants will be recruited in the Paris region.

SUMMARY:
Linguistic irregularities in number naming systems, such as the inversion of number words, affect the processing of Arabic numerals. Recently, it has been claimed that there is even a syntactic representation of number words. participant investigate the neurofunctional correlates of the syntactic processing of number words by examining different levels of place-value processing in a study with two complementary successive phases (Group 1 and Group 2) in healthy adults. In the first phase with Group 1, participant evaluate the unit-decade compatibility effect (UDCE) in two-digit magnitude comparisons. In the second phase with Group 2, participant investigate the carry-over effect in two-digit addition problems.

DETAILED DESCRIPTION:
Selection visit

* Call for participants for pre-selection
* Sending of information forms by mail
* Making an appointment for the inclusion visit at GHU Paris
* Information on the modalities, constraints and foreseeable risks of the study
* Collection of informed consent
* Verification of inclusion/non-inclusion criteria
* Clinical examination:

  * Verification of medical history and drug treatments
  * Psychiatric pathology
  * Consumption of toxic substances (nicotine, alcohol, cannabis, etc.)
  * Manual lateralization will be assessed by the score on the Edinburgh questionnaire (Oldfield, 1971)
* Collection of main medical history and concomitant treatments
* Explanation of study procedures
* MRI examination

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 to 45 years;
* Female or male;
* Right-handed preference;
* Subject, or legal representative, who has given consent to participate;
* Native language: French
* Subject affiliated with a social security system;
* Having signed their consent to participate (and their legal representative if applicable),
* Subjects have read the information letter and given their free and informed consent;
* Normal medical, neurological, and neuroradiological examinations
* For women of childbearing age, be on effective contraception

Exclusion Criteria:

* Not corresponding to the targeted age range;
* Subject with contraindications to an MRI examination (pacemaker or neurosensory stimulator or implantable defibrillator, cochlear implants, ferromagnetic foreign bodies in the eyes or brain near neural structures, metal prostheses, patient agitation: non-cooperative or agitated patients, minors, claustrophobic subjects, pregnant women, ventriculoperitoneal neurosurgical shunt valves, dental braces);
* Subject with chronic alcohol or drug use;
* Abuse or dependence on substances (except nicotine) or toxic substances for more than 5 years or having led to comas (overdoses);
* Subject with sudden-onset cognitive disorders that could indicate a stroke; a history of head trauma with loss of consciousness for more than 1 hour, or encephalitis;
* Subject with chronic neurological, psychiatric, endocrine, hepatic, or infectious conditions;
* Subject with a history of major illness (diabetes, chronic lung disease, severe cardiac, metabolic, hematological, endocrine, or immunological disorder, cancer);
* Subject on medication: taking medications likely to interfere with brain imaging measurements (psychotropics, anxiolytic hypnotics, neuroleptics, anti-Parkinsonians, benzodiazepines, steroidal anti-inflammatories, antiepileptics, central analgesics, and muscle relaxants);
* Color blindness;
* Inability to comply with the study for geographical or psychiatric reasons;
* Tattoo incompatible with MRI;
* Cerebral palsy;
* Fine motor skills disorder;
* Pregnant women at the time of inclusion;
* Adult subjects under legal protection or unable to give consent (article L.1121-8 of the French Public Health Code) (under guardianship or curatorship);
* Children and parents under legal protection measures

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: In the experimental phase, 42 adult volunteers (a total of 84), selected according to strict criteria, will undergo an MRI scan, each comprising: - anatomical acquisition, - functional acquisition of activation during a number processing task (Phase 1: two-digit number magnitude comparison; Phase 2: multi-digit mental arithmetic).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Neurofunctional variables (fMRI) | Day 1
  the comparison of pairs of incompatible numbers compared to pairs of compatible numbers during the comparison of numbers.
Structural variables (structural MRI) | Day 1
  the comparison of problems of addition with and without restraint during mental arithmetic.
Behavioral variables, | Day 1
  we compare performance to the post-imaging reading test
structural variables | Day 1
  recording of morphological and brain morphometric characteristics.

SECONDARY OUTCOMES:
Handedness score | Day 1
  Measuring the lateralization of the hand will allow to recognize, based on the proposed activities, the dominant hand.
Demographics questionnaire | Day 1
  this questionnaire which will allow the collection of all the precise information about the participant

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Ste Anne, Paris, France